CLINICAL TRIAL: NCT01598324
Title: Functional and Neurochemical Correlates of Treatment Response in Major Depressive Disorder
Status: Terminated | Type: Observational
Why Stopped: Clinical trial from which subjects were recruited closed to enrollment
Sponsor: Mclean Hospital (Other)
Collaborators: Pfizer (Industry); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tara Lauriat, Principal Investigator, Mclean Hospital
Other Study IDs: WS2058787
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Treatment-Resistant Depression
Keywords: magnetic resonance imaging; magnetic resonance spectroscopy; depression; escitalopram; selective serotonin reuptake inhibitor; treatment-resistant depression; ziprasidone
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- escitalopram responders no augmentation: Participants who show a clinical response following 8 weeks on an SSRI will have a final magnetic resonance scan at the end of 8 weeks and will complete the study at that time.
- Ziprasidone augmentation: Participants who do not respond to escitalopram and are randomized to ziprasidone augmentation will have a final magnetic resonance scan following 8 weeks on ziprasidone.
- Placebo augmentation: Participants who do not respond to escitalopram and are randomized to placebo augmentation will have a final magnetic resonance scan following 8 weeks on placebo.

SUMMARY:
This is an ancillary study to a clinical trial that is being conducted at Massachusetts General Hospital. Investigators at MGH are conducting a clinical trial to test the efficacy of ziprasidone together with escitalopram for treatment-resistant depression (NCT00633399). This observational study will involve magnetic resonance scans to examine brain chemistry (neurotransmitter levels), brain activity, and functional connections between brain regions before and after participating in the trial. The neurotransmitters of interest are glutamate, glutamine, and GABA. Comparisons will be made between individuals who receive ziprasidone and individuals who receive an inactive placebo. Differences between participants who respond to standard antidepressants and those who require additional medication will also be examined. All participants will have a baseline magnetic resonance scan before starting medication. The second scan will be after 8 weeks of escitalopram treatment for those who respond or following 8 weeks of escitalopram plus ziaprasidone or placebo (16 weeks after starting) for those who do not respond to escitalopram alone. Participants will complete standard rating scales for depression at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Meets DSM-IV criteria for major depressive disorder
* Meets eligibility criteria for clinical trial of ziprasidone augmentation of escitalopram
* Capable of providing informed consent

Exclusion Criteria:

* Meets exclusion criteria for augmentation clinical trial protocol
* Pregnancy or unwillingness to avoid pregnancy during trial
* Current or past psychosis or bipolar disorder
* Substance abuse or dependence in the past six months
* Clinically significant suicidality
* Unstable cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease or uncontrolled seizures
* Use of a concomitant medication that acts on glutamate or GABA neurotransmission
* Contraindication to magnetic resonance imaging (metal implant or device, occupational metal exposure, significant claustrophobia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in a clinical trial for treatment-resistant depression who agree to have magnetic resonance scans
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Glutamate level in antidepressant non-responders | 8 weeks after starting combination therapy phase
  Glutamate levels are measured by magnetic resonance spectroscopy 8 weeks after starting treatment with ziprasidone or placebo in addition to escitalopram.

SECONDARY OUTCOMES:
Glutamine level in treatment-responders following six weeks of antidepressant and non-responders following six weeks of adjunctive treatment. | 8 weeks or 16 weeks
Glutamine level in treatment-responders following six weeks of antidepressant and non-responders following six weeks of adjunctive treatment | 8 weeks
GABA level in treatment-responders following six weeks of antidepressant and non-responders following six weeks of adjunctive treatment | 8 weeks
Glutamine level in antidepressant non-responders | 8 weeks
  Glutamine levels are measured by magnetic resonance spectroscopy 6 weeks after starting treatment with ziprasidone or placebo together with escitalopram.
GABA level in antidepressant non-responders | 8 weeks
  GABA levels are measured by magnetic resonance spectroscopy 6 weeks after starting treatment with ziprasidone or placebo together with escitalopram.
Functional connectivity in default mode network measured by functional magnetic resonance imaging (fMRI) in treatment-resistant individuals receiving adjunctive treatment | 8 weeks after starting combination therapy phase
  Functional connectivity will be measured by performing fMRI in the resting state.
Functional connectivity in default mode network measured by functional magnetic resonance imaging (fMRI) in treatment-resistant individuals receiving adjunctive treatment and treatment-responders receiving an antidepressant | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital - McLean Imaging Center, Belmont, Massachusetts, United States